CLINICAL TRIAL: NCT06034184
Title: To Evaluate Whether Virtual Reality Compared to Standard Education Improves Nursing Students' Ability to Triage in a Simulated Mass Casualty Incident- a RCT
Brief Title: Enhancing Mass Casualty Triage Through Virtual Reality Simulation
Acronym: VR-MCI-RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sophiahemmet University (Other)
Collaborators: Falck Ambulance A/S (Unknown); CrashCourse AB (Unknown)
Responsible Party: Principal Investigator, Veronica Lindström, Professor and Registered Nurse, Sophiahemmet University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EPM:2023-02154-02
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Learning; Mass Casualty Incident; Triage; Training
Keywords: Virtual Reality; Mass casualty incidents; Triage; Learning; Nursing Students

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Using Virtual Reality for training and learning mass casualty incidents (Experimental): The nursing students use glasses and handcontrollers (High Fidelity Simulation) in the VR scenario for training and learning mass casualty incidents.
  Interventions: Other: Virtual Reality
- Standard education and training (No Intervention): Standard education, including lectures and paper exercises

INTERVENTIONS:
Other: Virtual Reality — The nursing students use glasses and handcontrollers (High Fidelity Simulation) in the VR scenario for training and learning mass casualty incidents.
  Other Names: Training mass casualty incidents
  Arms: Using Virtual Reality for training and learning mass casualty incidents

SUMMARY:
This interventional study aims to investigate whether Virtual Reality (VR) compared to traditional education and training, can enhance the correct triage abilities of nursing students in simulated mass casualty incidents (MCI). The primary research question seeks to answer if VR compared to Standard education supports students' ability to triage correctly in a simulated MCI situation. Additionally, this study aims to address the following secondary questions: Does VR compared to standard education have an effect on the time to triage in a simulated MCI situation? And, does VR compared to Standard education have an effect on theoretical knowledge retention concerning triage in MCI situations? In the interventional group, participants will utilize VR for MCI training and learning, while the control group will undergo standard education, including lectures and paper exercises. The researchers will compare the two groups of nursing students to assess whether VR yields better outcomes in MCI triage education.

DETAILED DESCRIPTION:
A randomized controlled trial (RCT) involving nursing students from a university in Stockholm, Sweden. The students are randomly allocated in a 1:1 ratio to either VR (intervention) or standard training in triaging during a mass casualty Incident. Both groups of participants will receive the same lecture on disaster events and triage using the same method before undergoing triage training either with VR support or traditional paper-based training. To achieve a power of 0.80 and a p-value of 0.05, a total of 60 participants are required (control n=30, intervention n=30). However, all students (approximately 100) will be invited to participate in the study to avoid excluding those who wish to take part in the study. The primary outcome measure is the students' ability to triage correctly. Secondary outcome measures include knowledge and knowledge retention, as well as the time taken to triage correctly. Knowledge tests will be conducted approximately one week after training and again 3-6 months after completing the training. The knowledge test consists of a questionnaire with 20 multiple-choice questions used in previous studies.

ELIGIBILITY:
Inclusion Criteria:

Nursing students registered for a course in disaster medicine/emergency care that is conducted during their fifth semester (out of 6) in the nursing program.

Exclusion Criteria:

Does not meet inclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants performing correct triage | From enrollment, theoretical education and performing training on mass casualty incidents with or without Virtual Reality
  Measuring if VR compared to Standard education has an effect on the frequency of correctly triage

SECONDARY OUTCOMES:
Time range on performing correct triage on 10 injured | From enrollment, theoretical education and performing training on mass casualty incidents with or without Virtual Reality
  Measuring if VR compared to Standard education has an effect on the time to triage correctly (10 patients) in a simulated MCI situation

OTHER OUTCOMES:
Number of participants with correct answers in theoretical tests | From enrollment, the training on mass casualty incidents with or without Virtual Reality and measuring nursing students theoretical knowledge retention on triage 1 week- 3-6 months after training.
  To measure if VR compared to Standard education has an effect on theoretical knowledge retention

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Lindström, PhD, Principal Investigator — Sophiahemmet University
Locations (1):
- Sophiahemmet University, Lindstedtvägen 8, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
The data analyzed and presented will be available from the PI and/or corresponding author (when published) on reasonable request